CLINICAL TRIAL: NCT00825331
Title: Improvement of Periprocedural Guidewire Management for Cardiac Catheterization (PTCA)Using Preprocedural Marking of the Arterial Access Site and a Graduated Scheme for Removal of the Guidewire
Brief Title: Improvement of Periprocedural Guidewire Management for Cardiac Catheterization (PTCA)
Status: Withdrawn | Type: Observational
Why Stopped: Change of location for Investigators
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Other Study IDs: Guidewire Management for PTCA
Record Dates: First submitted 2009-01-19; First posted 2009-01-21 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Cardiac Catheterization
Keywords: guide wire; cardiac catheterization; ultrasound-guided examination of the access site; graduated scheme; elective and non elective cardiac catheterization

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: patients for elective catheterization without special risks
- 2: patients for elective catheterization with special risks
- 3: patients for PCI without GP IIb/IIIa
- 4: Patients for PCI with GPIIb/IIIa and emergencies

SUMMARY:
Periprocedural management of guidewire placement and removal in patients needing cardiac catheterization by use of marking of the access site and removal procedure due to a graduated scheme

DETAILED DESCRIPTION:
Before elective cardiac catheterization, patients undergo an ultrasound-guided marking of the bifurcation of the common femoral artery in order to access the vascular complication rate compared tho those of non-marked patients.

Concerning the removal of the guided wire, patients will be treated due to a graduated scheme taking care of different risk levels. This procedure should improve clinical routine, but the efficacy and safety have to be assessed. Depending on the risk level, the guide wire will be removed either by an ambulance officer or emergency medical technician, assistant personal of the cardiac catheterization operating room or by a physician specialist in intensive care. Both methods should lead to quality assurance.

ELIGIBILITY:
Inclusion Criteria:

* elective cardiac catheterization or PCI or emergency interventions

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients needing elective cardiac catheterization or PCI or emergency interventions
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Decrease of vascular complications by marking of the access site | 18 months

SECONDARY OUTCOMES:
Improvement of guide wire removal procedure by using the graduated scheme | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Emilia Stegemann, MD, Principal Investigator — RWTH Aachen University Departement of Cardiology, Pulmonology and Vascular Medicine
Locations (1):
- Department of Medicine, Division of Cardiology, Pulmonology and Vascular Medicine, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Stegemann E, Busch L, Stegemann B, Lauer T, Hoffmann R, Heiss C, Kelm M. Evaluation of a structured training program for arterial femoral sheath removal after percutaneous arterial catheter procedures by assistant personnel. Am J Cardiol. 2015 Apr 1;115(7):879-83. doi: 10.1016/j.amjcard.2015.01.012. Epub 2015 Jan 15. PMID 25661570